CLINICAL TRIAL: NCT03600129
Title: Ultrasound-guided Quadratus Lumborum Block for Postoperative Pain Control After Endoscopic Prostatectomy - Double Blinded, Placebo-controlled, Randomised Trial.
Brief Title: Qudratus Lumborum Block for Postoperative Pain After Endoscopic Prostatectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bartosz Horosz, MD, MD, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 83/PB/2018
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: regional anesthesia; quadratus lumborum block; patient controlled anesthesia; laparoscopic prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, randomised
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Solution used for block (local anesthetic or placebo) is known to anesthetist not involved in patient's care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB with 0,375% ropivacaine (Experimental)
  Interventions: Procedure: Qadratus Lumborum Block; Drug: 30 milliliters of 0.375% Ropivacaine
- QLB with 0,9% NaCl (Placebo Comparator)
  Interventions: Procedure: Qadratus Lumborum Block; Drug: 30 milliliters of 0.9% NaCl

INTERVENTIONS:
Procedure: Qadratus Lumborum Block — Bilateral, ultrasound - guided Quadratus Lumborum Block
Drug: 30 milliliters of 0.375% Ropivacaine — 30 milliliters of 0.375% Ropivacaine used for Quadratus Lumborum Block
  Arms: QLB with 0,375% ropivacaine
Drug: 30 milliliters of 0.9% NaCl — 30 milliliters of 0.9% NaCl used for Quadratus Lumborum Block
  Arms: QLB with 0,9% NaCl

SUMMARY:
Laparoscopic prostatectomy (LP) is characterized by substantial tissue trauma, despite its minimally -invasive approach. Although postoperative pain intensity is lower when compared to open procedures, the use of opioids is common. Retrospective review of available LP cases revealed that although analgesic demand varied, nearly all of our LP patients required opioids postoperatively. Bilateral Quadratus Lumborum Block (QLB), being one of relatively new features of regional anesthesia, offers good analgesia of abdominal wall, with the potential for control of visceral pain. This study was established to evaluate its effectiveness in alleviating pain after radical prostatectomy in a double - blind, placebo - controlled manner.

ELIGIBILITY:
Inclusion Criteria:

* ASA status less or equal 3
* Scheduled for transperitoneal or extraperitoneal endoscopic prostatectomy
* Able to understand information provided and to sign the informed consent for participation in the study

Exclusion Criteria:

* known allergy to local anesthetics and opioids
* infection in the area of block placement
* known chronic use of opioids, gabapentinoids and tricyclic antidepressants
* mental inability to understand the principles and rules of patient-controlled analgesia pump

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Opioid consumption following prostatectomy | 24 hours
  Oxycodone consumption with Patient-Controlled Analgesia pump

SECONDARY OUTCOMES:
Pain score | 24 hours
  Pain scores assessed with Numeric Rating Scale (NRS).In this scale pain intensity is expressed using one of the numbers 0 - 10, 0 being no pain and 10 worst pain imaginable.
Time to first dose of opioid | 24 hours
  Time in minutes from emergence from anesthesia to the first request for opioid
Opioids - related complications | 24 hours
  The occurence of symptoms and conditions related to the use of opioids, like nausea, ileus, itching

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Malec-Milewska, MD, PhD, Study Chair — Orlowski Hospital, Centre of Postgraduate Medical Education, Department of Anesthesiology and Intensive Care
Locations (1):
- Centre of Postgraduate Medical Education,Department of Anesthesia and Intensive Care, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No